# Using Social Media to Decrease Healthcare Utilization for Pediatric Asthma: a Pilot Randomized Control Trial

NCT05013788

Version Date: 07/28/2021

Contact Name: Dr. Raymond Parlar-Chun Telephone:



#### PARENTAL PERMISSION TO TAKE PART IN RESEARCH

**Study Title:** Social Media for Pediatric Asthma

Protocol No.: HSC-MS-21-0426

Principal Investigator: Raymond Parlar-Chun, Pediatrics, UTHealth

We are doing this research study to learn more about how social media can be used to provide you and your child with ongoing asthma education to help decrease the need for hospitalization, ER visits, or clinic visits for asthma. You are being invited to be in this research study because your child has been hospitalized for asthma. Please feel free to ask questions at any time. Your participation is voluntary and you can stop at any time without penalty. Your participation will not affect the care your child is receiving currently.

If you agree to participate in this study:

- We will collect information from your child's medical records. We will collect information about the frequency and cost of your child's hospitalization, emergency room visit, or clinic visits within one year of enrollment.
- Each month (12 phone follow ups) we will contact you to determine if your child had been hospitalized, visited the ER, or visited the clinic within that month as well as a brief survey. We anticipate the phone calls taking no more than 10 minutes. You do not have to answer any questions that you do not wish to answer.
- If you are part of the intervention group, you will be asked to join our social media accounts on Facebook, Twitter, SnapChat, and/or Instagram. We will use these platforms to provide education to you and/or your child. No personal health information will be shared on these sites.

If you successfully complete the 12 follow up phone follow ups, you will be awarded a \$50 gift card at the end of one year.

Every research study involves some risk to your confidentiality. It's possible that other people could find out you and your child were in the study or see your child's study information. But we will take every step to keep this from happening, so we think this risk is very low. We don't know if you and your child will benefit from being in this study. However, we hope the results of this study will help improve asthma education for families that have children with asthma.

The identifiable information (e.g., your child's name, medical record number, or date of birth) or collected in this study will NOT be used or shared for future research studies, even if we remove the identifiable information like your child's name, medical record number, or date of birth.

Contact Name: Dr. Raymond Parlar-Chun Telephone:

IRB NUMBER: HSC-MS-21-0426
UTHealth
The University of Texas

### **Parental Permission Social Media for Pediatric Asthma**

I am happy to answer any questions you may have about this research study. If you have questions about your rights as a research participant, or if you have any concerns, comments, or complaints related to participating in this study, please contact the UTHealth Institutional Review Board at

If you sign this document, you give permission to UTHealth and Memorial Hermann Health System to use and disclose (release) your child's health information. The health information that we may use or disclose for this research includes the frequency and cost of your child's hospitalization(s), emergency room visit(s), or clinic visits within one year of enrollment. Please understand that health information used and disclosed may include information relating to HIV infection, drug abuse, alcohol abuse, behavioral health, and psychiatric care.

People who receive your child's health information may not be required by Federal privacy laws (such as the Privacy Rule) to protect your child's health information and may share your child's information with others without your permission, if permitted by laws governing them. Your child will not be personally identified in any reports or publications that may result from this study. If all information that does or can identify your child is removed from your child's health information, the remaining information will no longer be subject to this authorization and may be used or disclosed for other purposes.

Representatives of UTHealth and Memorial Hermann Health System will see your child's name and other personal identifiers when they review your child's research records and medical records for the purposes of verifying study data.

Please note that you do not have to sign this Authorization, but if you do not, your child may not participate in this research study. UTHealth and Memorial Hermann Health System may not withhold treatment or refuse treating your child if you do not sign this Authorization.

You may change your mind and revoke (take back) this Authorization at any time. Even if you revoke this Authorization, researchers may still use or disclose health information they already have obtained about your child as necessary to maintain the integrity or reliability of the current research. To revoke this Authorization, you must contact Dr. Raymond Parlar-Chun in writing at

This Authorization will expire 6 years after the end of the study.

If your child will reach the legal age of majority (18 in the state of Texas) and is able to provide his or her own consent while enrolled as a participant in this study, the study team will contact him or her to obtain his or her adult consent.

Contact Name: Dr. Raymond Parlar-Chun Telephone:



IRB NUMBER: HSC-MS-21-0426 UTHealth IRB APPROVAL DATE: 07/28/2021

## Parental Permission Social Media for Pediatric Asthma

Page 3

### **SIGNATURES**

| Sign below only if you understand the information given to you about the research and you choose to |
|---|
| take part in this research study. Make sure that all your questions have been answered. If you decide to |
| take part in this research study, a copy of this signed consent form will be given to you. |

| Printed Name of Participant | | | |
|---|---|---|---|
| Printed Name of Parent or<br>Guardian | Signature of Parent or Guardian | Date | Time |
| Printed Name of Person Obtaining Informed Consent | Signature of Person Obtaining Informed Consent | Date | Time |

Contact Name: Dr. Raymond Parlar-Chun Telephone:

